CLINICAL TRIAL: NCT00851682
Title: Feasibility Study of Prostate Tumor Localization for Focal Cryoablation of Prostate Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was stopped and will not resume. Participants are no longer being examined.
Sponsor: Washington University School of Medicine (Other)
Collaborators: Midwest Stone Institute. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: HRPO#03-0535
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Results first posted 2015-11-11 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Dynamic Contrast Enhanced MRI; Non-invasive Prostate Cancer Detection
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radical prostatectomy patients (Other): Patients who have been diagnosed with prostate cancer and are scheduled to undergo radical prostatectomy and have not received any preoperative treatment for prostate cancer.
  Interventions: Device: MRI scan
- Brachytherapy patients (Other): Patients who have been diagnosed with prostate cancer and are scheduled to undergo brachytherapy and have not received any preoperative treatment for prostate cancer.
  Interventions: Device: MRI scan

INTERVENTIONS:
Device: MRI scan — Each patient will undergo one, contrast-enhanced MRI scan prior to his planned, standard of care procedure, either radical prostatectomy or brachytherapy, depending on the study arm. Patients will be randomized to be imaged with either a phased array body coil or an endorectal coil.

SUMMARY:
The purpose of the present study is to find out if MRI techniques examining (1) the motion of water molecules in the prostate (diffusion sensitive MRI), (2) the difference in blood flow to the prostate (dynamic contrast enhanced MRI), and (3) differences in chemical composition of the prostate (MR spectroscopy), can be used to detect prostate cancer early and non-invasively. Localization of the cancer within the prostate would be of particular importance in focal cryoablation of prostate carcinoma which we hope to improve as a result of this project.

Additional aim of the study is to correlate expression of genes believed to pay a role in prostate cancer with MRI findings.

DETAILED DESCRIPTION:
Radical prostatectomy patients will undergo an MRI prior to their scheduled surgery. Ex vivo imaging will be done on prostates once removed. Results from the final pathology with be compared with results of imaging to determine the accuracy of the image analysis in cancer localization and staging.

Brachytherapy patients will undergo an MRI prior to their scheduled procedure. Two areas of suspected cancer and two areas without suspected cancer will be prospectively identified based on the MRI imaging. At the time of brachytherapy, transrectal needle biopsies will be obtained from the previously identified areas. The needle cores will be reviewed by study pathologist to determine the accuracy of the image analysis in cancer localization and staging.

ELIGIBILITY:
Inclusion Criteria:

* patients who have been diagnosed with prostate cancer and are scheduled for radical prostatectomy or for brachytherapy
* patients who have not received any preoperative treatment for their diagnosis of prostate cancer

Exclusion Criteria:

* patients with implants that are electronically, magnetically, or mechanically active
* patients with intracranial aneurysm clips
* patients who have undergone cosmetic eyelid surgery
* patients with history of pheochromocytoma, insulinoma and acute glaucoma
* patients with estimated glomerular filtration rate (eGFR) less than 60 ml/min/1.73m2

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2009-01; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Grubb, III, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radical Prostatectomy Patients | Brachytherapy Patients
Started | 60 | 5
Completed | 55 | 5
Not Completed | 5 | 0
Not completed — screen failure | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radical Prostatectomy Patients | Brachytherapy Patients | Total
Number analyzed (Participants) | 60 | 5 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 2 | 43
  >=65 years | 19 | 3 | 22
Age, Continuous [Mean (Full Range); unit: years] | 60 [39 to 76] | 66 [58 to 73] | 61 [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 60 | 5 | 65
Region of Enrollment [Number; unit: participants]
  United States | 60 | 5 | 65

OUTCOME MEASURES:

1. Primary Outcome: Improved Accuracy of Prostate Cancer Detection by MRI Scan.
Description: Data obtained as part of this study could not be analyzed in a meaningful way due to problems with correlation between the cancerous tissue identified by histology and tissue imaging from imaging.
Time Frame: At time of treatment
Population: Data obtained as part of this study could not be analyzed in a meaningful way due to problems with correlation between the cancerous tissue identified by histology and tissue imaging from imaging.
Arm/Group | Radical Prostatectomy Patients | Brachytherapy Patients
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Successful MRI Guidance of Transrectal Ultrasound Biopsy in Patients.
Description: Ultrasound guidance of transrectal ultrasound biopsy was not attempted.
Time Frame: At time of treatment
Population: as for outcome 1
Arm/Group | Radical Prostatectomy Patients | Brachytherapy Patients
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Radical Prostatectomy Patients | Brachytherapy Patients
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/5
Other Adverse Events (participants affected / at risk) | 0/60 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes